CLINICAL TRIAL: NCT06783140
Title: Comparing Second-Line NABPLAGEM vs. Nab-paclitaxel/Gemcitabine in BRCA1/2 or PALB2 Mutant Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Study of NABPLAGEM vs. Nab-Paclitaxel/Gemcitabine in BRCA1/2 or PALB2 Pancreatic Cancer
Acronym: PLATINUM-CAN
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLATINUM-CAN; CAPCR 24-5124 (Other: University Health Network)
Record Dates: First submitted 2025-01-16; First posted 2025-01-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer, Advanced or Metastatic; BRCA1/2 Mutation; PALB2 Gene Mutation
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Taxes; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1- NABPLAGEM (Nab-paclitaxel+Cisplatin+Gemcitabine) (Experimental): Nab-paclitaxel 100 mg/m2 + cisplatin 25 mg/m2 + gemcitabine 800 mg/m2 on days 1 and 15 of every cycle.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine; Drug: Cisplatin
- Arm 2 - Nab-paclitaxel+gemcitabine (Active Comparator): Nab-paclitaxel 125 mg/m2 + gemcitabine 1000 mg/m2 on days 1 and 15 of every cycle.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nab paclitaxel — Paclitaxel Powder For Injectable Suspension Nanoparticle, Albumin-bound Paclitaxel is an albumin-stabilized nanoparticle formulation of the natural taxane paclitaxel with antineoplastic activity.
Drug: Gemcitabine — Gemcitabine is a hydrochloride salt of an analogue of the antimetabolite nucleoside deoxycytidine with antineoplastic activity.
Drug: Cisplatin — Cisplatin is an alkylating-like inorganic platinum agent (cis-diamminedichloroplatinum) with antineoplastic activity.
  Arms: Arm 1- NABPLAGEM (Nab-paclitaxel+Cisplatin+Gemcitabine)

SUMMARY:
This study will compare two different regimens for patients with BRCA1/2 or PALB2 mutated metastatic pancreatic cancer after progression on first-line FOLFIRINOX.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic adenocarcinoma. Adenosquamous carcinoma, squamous carcinoma, acinar cell carcinoma, and carcinoma not otherwise specified are also acceptable.
* BRCA1/2 or PALB2 mutation (somatic or germline).
* Measurable disease.
* Potential trial participants should have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment.
* Clinical or radiographic progression on first-line FOLFIRINOX (or NALIRIFOX) for metastatic disease.

  * Patients whose front-line chemotherapy was required to be simplified due to toxicity associated with any of the constituent components of FOLFIRINOX/NALIRIFOX (e.g. simplified to FOLFOX, FOLFIRI, 5-FU (including capecitabine)) will be eligible.
  * Patients with progressive disease while on maintenance PARP inhibitor treatment after FOLFIRINOX (or NALIRIFOX), irrespective of how long ago they received FOLFIRINOX/NALIRIFOX, will also be eligible.
  * Patients who develop metastatic disease during or within 6 months after completing FOLFIRINOX/NALIRIFOX in either the locally advanced or adjuvant/neoadjuvant settings will be eligible.
* Age 18 years or older.
* Ability to understand and willing to sign a written informed consent document.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 (Karnofsky Performance Status ≥60).
* Required Initial Laboratory Values
* Not pregnant and not nursing.

Exclusion Criteria:

* Patients may not have received prior cisplatin for their pancreatic cancer in any setting.
* Patients with > grade 2 peripheral sensory neuropathy are not eligible.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for at least 8-weeks. Patients with known, new or progressive brain metastases (active brain metastases) or leptomeningeal disease are ineligible.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load anytime within 6 months prior to registration are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Concomitant Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study. Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2031-06-02 (Estimated); Study Completion 2031-06-02 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 12 months
  The proportion of patients who achieve complete response (CR) or partial response (PR)
Overall Survival (OS) Time | 6 years
  The time form the date of randomization to the date of death

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 6 years
  Time from the date of randomization to the date of first documented disease progression or death
Duration of Response (DoR) | 6 years
  The time that criteria are met for complete response (CR) or partial response (PR) until the first date that recurrence or disease progression is objectively documented.
CA19-9 Response | 6 years
  Percentage decrease in CA19-9
Number of Adverse Events | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Erica S Tsang, MD, Principal Investigator — Princess Margaret Cancer Centre/University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada